CLINICAL TRIAL: NCT05967520
Title: A Phase IIa ,Randomized, Double-blind, Placebo-controlled, Dose-exploration Study of JMKX000189 in Treatment of Moderate to Severe Active Systemic Lupus Erythematosus
Brief Title: JMKX000189 for Moderate to Severe Active Systemic Lupus Erythematosus
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jemincare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: JY-R105-201
Record Dates: First submitted 2023-07-21; First posted 2023-08-01 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-10

CONDITIONS: Lupus Erythematosus, Systemic
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- JMKX000189 - higher dose (Experimental): Randomized 16 patients will be received JMKX000189 at a higher dose in oral continuously from Week 0 to Week 12 in addition to SOC.
  Interventions: Drug: JMKX000189
- JMKX000189 - lower dose (Experimental): Randomized 16 patients will be received JMKX000189 at a lower dose in oral continuously from Week 0 to Week 12 in addition to SOC.
  Interventions: Drug: JMKX000189
- Placebo (Placebo Comparator): Randomized 16 patients will be received Placebo in oral continuously from Week 0 to Week 12 in addition to SOC.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: JMKX000189 — JMKX000189 will be administered orally once a day
  Arms: JMKX000189 - higher dose; JMKX000189 - lower dose
Drug: Placebo — Placebo will be administered orally once a day
  Arms: Placebo

SUMMARY:
The trial will evaluate pharmacodynamics，pharmacokinetics，safety，and efficacy of JMKX000189 versus placebo in participants with moderately to severely active systemic lupus erythematosus (SLE) while receiving standard of care (SOC) treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must have been diagnosed with systemic lupus erythematosus at least 24 weeks prior to screening and must be assessed to meet 2019 EULAR/ACR SLE classification criteria during screening.
2. the subject must meet one of the following at screening: a. ANA titer ≥1:80;b. anti-dsDNA antibody positive; c. Anti-Smith antibody positive.
3. At least one of the following SLE background standard therapies (including no more than one immunosuppressant) was required for 12 weeks prior to randomization, and the dose must remain stable at least 30 days until randomization and throughout study participation.

Exclusion Criteria:

1. Active lupus nephritis (defined as urinary protein >1g/24 h or urinary total protein/creatinine ratio (UPCR) >1 mg/mg (113 mg/mmol) within 8 weeks prior to screening or at randomization).
2. Active lupus of the central nervous system (CNS) (including epilepsy, psychosis, organic encephalopathy syndrome, cerebrovascular accident, encephalitis, or CNS vasculitis) within 60 days prior to randomization.
3. Myocardial infarction, unstable angina pectoris, stroke, transient ischemic attack, decompensated heart failure requiring hospitalization, grade III/IV heart failure, or untreated severe sleep apnea occurred ≤6 months before screening.
4. Previous or current atrioventricular block of degree Ⅱ or Ⅲ, sick sinus syndrome, symptomatic bradycardia, atrial flutter or atrial fibrillation, ventricular arrhythmia or syncope associated with heart disease, or other arrhythmia deemed clinically significant and requiring intervention or treatment.
5. A history of severe respiratory disease or interstitial pneumonia or pulmonary fibrosis，which were found by the medical history or lung function test or chest CT examination conducted during screening or within 3 months prior to screening;Or abnormal pulmonary function of medical significance: 1 second forced expiratory volume (FEV1) or forced vital capacity (FVC)<70% of the expected value, or FEV1 /FVC < 0.7.
6. Patients with significant abnormalities in liver, renal function and blood routine during screening, including glutamate aminotransferase (ALT) or aspartate aminotransferase (AST) exceeding 2 times the upper limit of normal value;Serum creatinine greater than 1.5 times the upper limit of normal;Hemoglobin <90g/L;White blood cell count <2.5×109/L, platelet count (PLT) <75×109/L;Lymphocyte count <0.8×109/L;Abnormal results of other laboratory tests may affect the completion of the test or interfere with the test results according to the investigator.
7. Use of cyclosporine, tacrolimus, pimelimus, and sirolimus within 1 month prior to randomization.
8. Use of thalidomide or lenalidomide within 2 months prior to randomization.
9. Rituximab, telitacicept, or leflunomide were used in the 6 months prior to randomization.
10. Use of Belliumab within 3 months prior to randomization.
11. Intravenous treatment with cyclophosphamide was received within 6 months prior to randomization or oral treatment with cyclophosphamide within 30 days prior to initial administration.
12. History of type 1 diabetes mellitus, or uncontrolled Type 2 diabetes mellitus with HbA1c> 8%, or diabetic subjects with organ involvement (e.g. retinopathy or kidney disease).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-09-21 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in Total Lymphocyte Count From Baseline to Week 12 | Baseline,Week 12

SECONDARY OUTCOMES:
Change from baseline to Week 4,8,12 and 16 in the modified SLEDAI (mSLEDAI) score | Baseline, Week 4, 8,12, and 16
Percentage of Participants Achieving a Systemic Lupus Erythematosus Responder Index-4 (SRI-4) Response at Week 4,8,12 and 16 | Baseline, Week 4, 8,12, and 16
Percentage of Participants Achieving No worsening in Physician Global Assessment (PGA) of Disease Activity at Week 4,8,12 and 16, No worsening defined as an increase of PGA < 0.3 Points from baseline | Baseline, Week 4, 8,12, and 16

CONTACTS AND LOCATIONS:
Overall Officials: Xiaofeng Zeng, Principal Investigator — Peking Union Medical College Hospital
Locations (17):
- China (17):
  - The First Affiliated Hospital of Bengbu Medical College, Bengbu, Anhui
  - Xuanwu Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - The First Affiliated Hospital of Henan University of science and Technology, Luoyang, Henan
  - Xinxiang Central Hospital, Xinxiang, Henan
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - Pingxiang People's Hospital, Pingxiang, Jiangxi
  - China-Japan Union Hospital of Jilin University, Changchun, Jilin
  - Binzhou Medical University Hospital, Binzhou, Shandong
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Jining First People's Hospital, Jining, Shandong
  - Huashan Hospital Affiliated to Fudan University, Shanghai, Shanghai Municipality
  - Renji Hospital Affiliated to Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Shanxi Bethune Hospital, Taiyuan, Shanxi
  - West China Hospital Sichuan University, Chengdu, Sichuan

IPD SHARING:
Plan to Share IPD: No